CLINICAL TRIAL: NCT06605339
Title: Virtual Reality on Pain, Fear and Emotional Experience During Port Needle Insertion in Pediatric Hematology and Oncology Patients
Brief Title: Virtual Reality on Pain, Fear and Emotional Experience During Port Needle Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Afyonkarahisar Health Science University (Unknown)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASBU portVR
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Cancer
Keywords: pediatric; cancer; virtual reality; pain; fear; emotional behavior
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The child in the control group did not receive any additional intervention.
- Virtual reality (Experimental): In the study, Oculus Quest 2 256 GB All-In-One Vr Virtual Reality Glasses were used, and the Epic Roller Coasters train game, an application that would attract the attention of children, was determined by the researchers. The virtual reality application was started 2 minutes before the procedure and continued until the procedure was completed.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — Virtual Reality Distraction
  Arms: Virtual reality

SUMMARY:
In pediatric hematology-oncology patients, the need for a central venous catheter may arise in some cases to provide treatment. Totally implanted vascular access devices are known as "ports," and port catheters are commonly used due to their lower risk of infection. To maintain the port system and prevent infection, the port needle should be replaced every 5-7 days. During the course of treatment, pediatric hematology-oncology patients undergo frequently repeated procedures associated with high levels of pain and distress. Pain and distress resulting from repeated procedures are often uncomfortable symptoms for pediatric patients and their families. There are pharmacological and non-pharmacological methods to reduce pain and anxiety during port needle procedures in pediatric hematology-oncology patients. One pharmacological method, distraction, increases pain tolerance by focusing attention away from the painful stimulus. This technique is used as a powerful tool for pain and anxiety management in pediatric pain. Virtual reality glasses, used as a distraction method, provide access to an interactive, three-dimensional, computer-simulated environment through a head-mounted device that blocks out real-world views. It is stated that distraction with virtual reality is a beneficial non-pharmacological method for children during hospital-based needle applications for pediatric patients. This study evaluated the effect of virtual reality on pain, fear, and emotional appearance related to needle procedures in pediatric hematology-oncology patients during port needle changes.

DETAILED DESCRIPTION:
The study was conducted at the Pediatric Hematology and Oncology Clinic of Afyonkarahisar Health Sciences University Health Practice and Research Center.

Research Hypotheses:

H1: There is a difference in pain and fear scores among patients who watch videos using virtual reality glasses during port needle changes.

H2: There is a difference in emotional appearance scores among patients who watch videos using virtual reality glasses during port needle changes.

Randomization:

A stratified randomization scheme was used for distributing the sample into groups. Stratification was done based on gender (female, male), age group (4-7, 8-12), and port duration (<1 month, >1 month).

Patients requiring port needle changes were assigned to groups according to the randomization scheme. No additional intervention was made for patients in the control group; they were observed during the procedure after obtaining consent. Patients in the study group were introduced to the virtual headset and informed that they could watch a video using the virtual reality headset during the procedure. The "Epic Roller Coasters" video game was initiated. If the child wanted to remove the glasses during the procedure, they were excluded from the study. Before the procedure, the fear score was determined by asking both the patient and the parent using the Children's Fear Scale. After the procedure, the pain levels were evaluated independently by the child, the mother, the attending nurse, and the researcher. Following the intervention, the child's emotional appearance was assessed by the nurse.

ELIGIBILITY:
Inclusion Criteria:

* The child having a port catheter in place.
* The child agreeing to voluntarily participate in the study.
* The parent agreeing to voluntarily participate in the study.
* Obtaining consent forms from both the child and the parent.

Exclusion Criteria:

The child had a physical or psychological deficits that would prevent the child from wearing the headset needed to watch virtual reality

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | after the port needle insertion
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10
Fear assesed by Child Fear Scale | after the port needle insertion
  The Child Fear Scale (CFS), this one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear.
emotional apperance assesed by Emotional Appearance Scale for Children | after the port needle insertion
  This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'.
  Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gulcin Ozalp Gerceker, Assoc. Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No